CLINICAL TRIAL: NCT02094781
Title: A Randomized, Double-blind, Placebo-controlled, Three-arm Trial to Evaluate the Effect of Using Whey Protein and Creatine Supplements on Muscular Strength in Weight-training Adult Males
Brief Title: Effect of Using Whey Protein and Creatine Supplements on Muscular Strength in Weight-training Adult Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 200616; RH01717 (Other: GSK)
Record Dates: First submitted 2014-02-27; First posted 2014-03-24 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Nutritional Status
MeSH Terms: interventions — Whey Proteins; Creatine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Whey protein and creatine supplement (Experimental): Each sachet contained 30g whey protein powder and 5g creatine powder, administered twice a day. The first serving was consumed with breakfast and the second serving was consumed within 60 minutes of completing training or in the evening on non-training days. Participants also drank at least 2 litres of water per day
  Interventions: Dietary Supplement: Whey protein and creatine supplement
- Whey protein only supplement (Active Comparator): Each sachet contained 30g of whey protein powder and 5g of bulking agent powder, administered twice a day. The first serving was consumed with breakfast and the second serving was consumed within 60 minutes of completing training or in the evening on non-training days. Participants also drank at least 2 litres of water per day
  Interventions: Dietary Supplement: Whey protein only supplement
- Placebo (Placebo Comparator): Each sachet contained 30g of isocaloric carbohydrate powder and 5g of bulking agent powder, administered twice a day. The first serving was consumed with breakfast and the second serving was consumed within 60 minutes of completing training or in the evening on non-training days. Participants also drank at least 2 litres of water per day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Whey protein and creatine supplement — Each sachet contained 30g whey protein powder and 5g creatine powder, administered twice a day. The first serving was consumed with breakfast and the second serving was consumed within 60 minutes of completing training or in the evening on non-training days. Participants also drank at least 2 litres of water per day
  Arms: Whey protein and creatine supplement
Dietary Supplement: Whey protein only supplement — Each sachet contained 30g of whey protein powder and 5g of bulking agent powder, administered twice a day. The first serving was consumed with breakfast and the second serving was consumed within 60 minutes of completing training or in the evening on non-training days. Participants also drank at least 2 litres of water per day
  Arms: Whey protein only supplement
Dietary Supplement: Placebo — Each sachet contained 30g of isocaloric carbohydrate powder and 5g of bulking agent powder, administered twice a day. The first serving was consumed with breakfast and the second serving was consumed within 60 minutes of completing training or in the evening on non-training days. Participants also drank at least 2 litres of water per day
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the effect of combined whey protein and creatine supplement, as compared with whey protein supplement alone, on change in upper and lower body strength.

ELIGIBILITY:
Inclusion Criteria:

* Recreationally active males
* Age 18 to 35 years
* BMI 19 to 29.9 kg/m2
* Weight training 3 to 4 times a week for at least 6 months before the trial

Exclusion Criteria:

* Participants with medical conditions including active heart disease, high blood pressure, renal or hepatic impairment type I or II diabetes, bipolar disease, pulmonary disease, thyroid disease, immune disorder, psychiatric disorder
* Dietary or herbal supplement used in the past 60 days to increase muscle mass
* Use of protein supplement in the past 7 days
* Use of thermogenic supplement or beverage in the past 7 days
* Use of Non-steroidal anti inflammatory drugs or corticosteroids in the past 7 days

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2013-12; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of combined whey protein and creatine supplement, as compared with whey protein supplement alone, on change in upper body strength from Baseline to Week 4. | Baseline, Week 2, 4, 8 and 12
  Body strength will be evaluated using Repetition maximum (1-RM) and bench and leg press exercise testing. 1-RM in weight training is the maximum amount of weight one can lift in a single repetition for a given exercise

SECONDARY OUTCOMES:
To evaluate the effect of combined whey protein and creatine supplement, as compared with whey protein supplement alone, on changes in upper and lower body strength from Baseline through Week 12 | Baseline, Week 2, 4, 8 and 12
  Body strength will be evaluated using 1-RM and bench and leg press exercise testing
To evaluate the effect of combined whey protein and creatine supplement, as compared with placebo, on changes in upper and lower body strength from Baseline through Week 12. | Baseline, Week 2, 4, 8 and 12
  Body strength will be evaluated using 1-RM and bench and leg press exercise testing
To compare changes in upper and lower body strength from Baseline through Week 12, between combined whey protein and creatine supplement, whey protein supplement alone, and placebo. | Baseline, Week 2, 4, 8 and 12
  Body strength will be evaluated using 1-RM and bench and leg press exercise testing
To compare changes in upper and lower body endurance from Baseline through Week 12, between combined whey protein and creatine supplement, whey protein supplement alone, and placebo. | Baseline, Week 2, 4, 8 and 12
  Body endurance will be measured using bench press and leg press exercise testing
To compare the changes in lean vs. fat body mass composition from Baseline to Week 12 between combined whey protein and creatine supplement, whey protein supplement alone, and placebo. | Baseline and Week 12
  Body composition [(fat-free mass and fat mass (grams and % body fat, bone mass)] will be calculated using Dual X-Ray Absorptiometry (DXA)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Miami, Florida, United States